CLINICAL TRIAL: NCT04103281
Title: Expression Profiles of Integrin αDβ2 on Neutrophils in Sepsis
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00033027
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis Patients
  Interventions: Other: Sepsis
- Control Patients

INTERVENTIONS:
Other: Sepsis — Sepsis patients in the ICU with a breathing tube
  Groups: Sepsis Patients

SUMMARY:
In this research study we want to learn more about the characteristics of neutrophils that are present in the blood and secretions from a breathing tube of patients with sepsis. Sepsis is a severe type of infection, affecting various parts of the body. Neutrophils are a type of white blood cell that are part of the body's immune system. Even though neutrophils are important in getting rid of germs, they also may be harmful to parts of the body by causing injury in the lungs in patients with sepsis. Neutrophils can change their character in sepsis. Because of this, it is important for doctors to know what kind of neutrophils are in the blood and secretions from the breathing tube of patients with sepsis so that they can work to develop therapies to prevent these cells from being harmful.

ELIGIBILITY:
Case Inclusion Criteria:

* sepsis patient in the ICU with a breathing tube

Control Inclusion Criteria:

* scheduled for an elective surgical procedure and need preoperative blood draw or will have an intravenous catheter placed for the purpose of their surgical procedure
* Plan to have endotracheal tube for planned procedures.

Exclusion Criteria:

* On chronic immunosuppressive drugs such as chronic corticosteroid use, or preexisting immunodeficiency diseases (oncology patients, patients with transplantation)

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from 2-50 years old at Boston Children's Hospital either in an ICU with sepsis or a healthy control coming for a surgical procedure.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neutrophil characteristics | One day
  measure and report β2 integrin expression on neutrophils from blood and tracheal aspirate between sepsis patients and non-sepsis patients in pediatric population

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States